CLINICAL TRIAL: NCT00697710
Title: A Phase Ib/IIa, Multiple-Dose, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of S-777469 in Subjects With Mild to Moderate Atopic Dermatitis
Brief Title: A Phase Ib/IIa, Double-Blind, Randomized Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of S-777469 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0710D1416
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — S-777469

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): 50 mg S-777469 or Placebo, BID
  Interventions: Drug: 50 mg S-777469; Drug: Placebo
- Cohort B (Experimental): 200 mg S-777469 or Placebo, BID
  Interventions: Drug: 200 mg S-777469; Drug: Placebo
- Cohort C (Experimental): 800 mg S-777469 or Placebo, BID
  Interventions: Drug: 800 mg S-777469; Drug: Placebo

INTERVENTIONS:
Drug: 50 mg S-777469 — S-777469, 50 mg BID
  Arms: Cohort A
Drug: 200 mg S-777469 — S-777469, 200 mg BID
  Arms: Cohort B
Drug: 800 mg S-777469 — S-777469, 800 mg BID
  Arms: Cohort C
Drug: Placebo — Matching Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled, sequential-cohort, dose-escalation study was to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of S-777469, a CB2 cannabinoid receptor agonist, in subjects with mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy males and females between 18 and 65 years of age at the time of obtaining the written informed consent
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent
* Subject satisfies the diagnostic criteria for mild to moderate atopic dermatitis (AD) as judged by the Physician's Global Assessment Score and modified criteria

All of these features must be present:

1. Pruritus
2. Eczema (acute, subacute, chronic) with the following characteristics:current or prior flexural lesions, lesions on the face, neck, and extensor surfaces, sparing of groin and axillary regions (no lesions)
3. History of a chronic and relapsing course of eczema
4. Personal or family history of atopy

   * Subject is judged to be in general good health based on medical history, physical examination, and routine laboratory tests performed at screen and baseline, with the exception of diagnosis of mild to moderate AD
   * Subject has a negative laboratory results for hepatitis B surface antigen, hepatitis C virus (anti-HCV antibodies), and Human Immunodeficiency Virus antibody screens
   * Female subjects have a negative pregnancy test at screen and baseline
   * Serum creatinine in the normal range [0.5 to 1.5 mg/dl]
   * Liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and gamma glutamyl transpeptidase [GGT]) within normal range
   * Negative screen for drugs of abuse at screen and baseline
   * Subject agrees to refrain from smoking for the duration of the trial
   * Subject has no clinically significant abnormality on screening or baseline electrocardiogram (ECG). Inclusion of a subject with any ECG abnormality at screening or baseline must be jointly agreed upon by both Study Investigator and Sponsor to be not clinically relevant within the context of the study, prior to enrollment
   * Use of adequate birth control, if of reproductive potential and sexually active Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 1 additional month after last administration/dose of study drug.

For females, adequate birth control methods will be defined as: oral contraceptives, intrauterine device or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam For males adequate birth control methods will be defined as double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam

* For female subjects, menopause is defined as one year without menses; if in question, a follicle-stimulating hormone of >40 U/ml must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable
* Subject has not used any topical or systemic treatments for AD for 3 weeks prior to the Day 1 visit (i.e., the washout period), including topical corticosteroids (3 weeks prior to the Day 1 visit), antihistamines (3 weeks prior to the Day 1 visit), herbal preparation, cosmetic or emollient preparations (3 weeks prior to the Day 1 visit), immunosuppressant drugs or corticosteroids (3 weeks prior to the Day 1 visit), any other AD treatments (including light treatment) for 3 weeks prior to the Day 1 visit
* Subject is willing to completely avoid the use of any prescription or nonprescription (including over the counter) drugs or any topical preparations [other than those topical emollient preparations provided by the study site during screening, e.g., Cetaphil® cream] for 3 weeks prior to the first dose of study drug and during the entire study
* If a subject does not discontinue all prior medications within 3 weeks of study start, he/she may be included in the study only if both the Study Investigator and Sponsor's Medical Monitor agree that this is not clinically relevant within the context of the study
* Use of hormone replacement therapy (for postmenopausal females) and/or use of oral, implantable, transdermal, or injectable contraceptive(s) will be allowed
* Subject is willing to avoid strenuous physical activity (i.e., strenuous or unaccustomed weight lifting, running, exercise, etc.) from the screening visit, throughout the study, and until the post-study follow-up visit
* Subject is willing to avoid grapefruit-containing products/medications for 72 hours prior to entry into the clinical research unit and for the duration of the study
* Subject has no history of frequent or recent acetaminophen use and is willing to refrain from use of acetaminophen throughout the trial and for 4 days after the last dose

Exclusion Criteria:

Subjects will not be eligible if they meet any of the following criteria:

* Subject is under the age of legal consent (see inclusion criteria), is mentally or legally incapacitated, has significant emotional problems at the time of study entry, or has a history of psychiatric disorders
* Active dermatologic conditions which may confound the diagnosis of AD, such as scabies, allergic contact dermatitis, seborrheic dermatitis, cutaneous lymphoma, ichthyosis, or psoriasis
* History of malignancy not in remission for >5 years
* Presence of comorbid conditions that would preclude participation in the study, including:

Immune compromised state, including recent chemotherapy, immunotherapy, or organ transplant History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal or urological History or clinical manifestations of significant neurological or psychiatric disorders Subject has an active, intercurrent infection Subject has a history of clinically significant hypersensitivity, anaphylaxis, or allergies to any drug compound In no circumstances should a subject who did not qualify under inclusion criteria regarding liver function tests (ALT, AST, and GGT) be re-screened and/or re-qualified for this study

* Subject has any acute or chronic condition or prior therapy that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study or otherwise would make the subject unsuitable for this study
* Subject has a history of drug abuse within 1 year prior to Day 1
* Subject consumes excess amounts of alcohol, defined as exceeding an average of 14 drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor, or any combination of them) within 2 months prior to Study Entry, or is unwilling to comply with the restricted use of alcohol from screening, throughout the study, and until study completion (post-study visit)
* Subject has used any systemic antibiotics for 3 weeks prior to the Day 1 visit (washout period)
* Subject is pregnant or lactating or intends to become pregnant or, in the case of a male subject, intends to father a child during the study period and for 1 month after the last dose of study medication
* Subject requires use of immunosuppressive drugs such as oral corticosteroids or inhaled corticosteroids
* Subject has donated blood within 6 weeks prior to Day 1 or plasma within 2 weeks prior to screening, or received blood products within 2 months prior to Day 1
* Subject has poor peripheral venous access
* Subject has participated in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to Day 1
* Any reason which, in the opinion of the investigator, interferes with the ability of the subject to participate to, or complete, the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | Throughout the study period
  Safety assessments included adverse event monitoring, vital sign measurements, physical examination measurements, 12-lead electrocardiograms assessments, and standard clinical laboratory safety tests (hematology, blood chemistry, and urinalysis).
Pharmacokinetic Assessments | Days 1, 7, and 14
  Pharmacokinetic endpoints included Cmax, Tmax, T1/2,12hr, T1/2,z, and AUC0-12h for each dose level of S-777469 based on the sampling schedule. Time to achieve steady state was determined for each dose level. Serum protein binding of S-777469 was determined for all cohorts. Plasma and urine concentrations of S-777469 was determined for single dose and multiple doses for all cohorts. The plasma and urine samples were used for determination of concentrations of metabolites of S-777469. Plasma and urine samples for single dose and multiple doses for Cohort B was used for metabolite profiling.

SECONDARY OUTCOMES:
Efficacy assessment: To assess the potential anti-pruritic and anti-inflammatory efficacy of S-777469 after single-dose administration and twice daily administration in subjects with mild-to-moderate Atopic Dermatitis | Change from baseline to Day 14
  The efficacy endpoints included Physician's Global Assessment, Patient Assessment of Pruritus (Visual Analog Scale), Subject Diary Cards, Itching Score, Severity Scoring Of Atopic Dermatitis Index for assessment of Eczema, Thymus And Activation-Regulated Chemokine Assessment, Digital Photography of AD lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States